CLINICAL TRIAL: NCT01178268
Title: XIENCE V Everolimus Eluting Coronary Stent System (EECSS) China: Post-Approval Randomized Control Trial (RCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-387
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Occlusion; Thrombosis (Stent Thrombosis); Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Drug eluting stents; Stents; Angioplasty
MeSH Terms: conditions — Coronary Occlusion; Thrombosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XIENCE V EECSS (Active Comparator): Patients who will receive this stent.
  Interventions: Device: XIENCE V EECSS
- CYPHER SELECT PLUS SECSS (Active Comparator): Patients who will receive this stent.
  Interventions: Device: CYPHER SELECT PLUS SECSS

INTERVENTIONS:
Device: XIENCE V EECSS — Patients who will receive this stent.
  Arms: XIENCE V EECSS
Device: CYPHER SELECT PLUS SECSS — Patients who will receive this stent.
  Arms: CYPHER SELECT PLUS SECSS

SUMMARY:
This is a prospective, randomized, active-controlled, open label, parallel two-arm, multi-center, post-approval study descriptively comparing the XIENCE V EECSS to the CYPHER SELECT PLUS Sirolimus-Eluting Coronary Stent System (SECSS) ("CYPHER SELECT PLUS") during commercial use in China.

DETAILED DESCRIPTION:
Objectives

* Confirm the safety and effectiveness of the XIENCE V EECSS for the treatment of patients in China
* Evaluate patient compliance with dual antiplatelet therapy (DAPT)
* Evaluate physician-determined XIENCE V EECSS acute performance, deliverability, and resource utilization

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria

  1. Patient must be at least 18 years of age
  2. The patient or patient's legally-authorized representative agrees to participate in this study by signing the Ethics Committee (EC)-approved ICF prior to procedure.
  3. Patient must agree to undergo all protocol-required follow-ups until the completion of his/her 2-year follow-up.
  4. Patient must not currently be and must agree not to become a participant in any other clinical trial until completion of his/her 2-year follow-up.

Angiographic Inclusion Criteria

1. Target lesion(s) must be located in a native de novo coronary artery with a visually estimated diameter between ≥ 2.25 and ≤ 4.0 mm.
2. Target lesion(s) must measure ≤ 28 mm in length by visual estimation.
3. A maximum of two de novo lesions can be treated, ie,

   1. One lesion in one vessel, OR
   2. One lesion in each of two vessels, OR
   3. Two lesions in one vessel

Exclusion Criteria:

* General Exclusion Criteria

  1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year post index procedure
  2. Patients with known renal insufficiency or failure (eg, serum creatinine level of > 2.5 mg/dL, or patient is on dialysis)
  3. Patient had an MI within 72 hours and creatine kinase-myocardial band isoenzyme (CK-MB) has not returned to the normal range at the index procedure
  4. Non-study PCI for lesions in a target vessel (including side branches) has been performed within 1 year prior to the index procedure
  5. Patient has a planned PCI (staged procedure) within 6 months from the date of the index procedure
  6. Left ventricular ejection fraction (LVEF) of < 30%.
  7. Any planned surgery necessitating discontinuation of antiplatelet therapy within 1 year
  8. Patient's current medical condition has a life expectancy of < 2 years
  9. Patient meets contraindications of the IFU

Angiographic Exclusion Criteria

1. Lesion located within an arterial or saphenous vein graft or distal to a diseased arterial or saphenous vein graft
2. Lesion located in left main coronary artery
3. Ostial lesion (within 3 mm of the aorta junction, or origin of the left anterior descending or left circumflex arteries)
4. Involves a bifurcation in which the side branch is ≥ 2 mm in diameter AND the ostium of the side branch is > 50% stenosed by visual estimation
5. Total occluded lesions (TIMI=0)
6. Restenotic lesions
7. Thrombus-containing vessel
8. Extreme angulation (≥ 90º) proximal to or within the lesion
9. Excessive tortuosity proximal to or within the lesion
10. Heavy calcification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gao Runlin, MD, FACC, Principal Investigator — Fu Wai Hospital
Locations (2):
- China (2):
  - Fu Wai Hospital, Beijing
  - Authorized Representative in China Guidant International Trading (Shanghai) Co., Ltd., Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 488 patients in the Per-protocol (PP) population for final analysis. First Patient Enrolled on August 18, 2010, Last Patient Enrolled on August 31, 2011 and the Final Database Lock was on September 26, 2013. The total patient enrollment rate was 0.5 patients/site/week based on 489 patients enrolled over 54 weeks at 20 sites.
Pre-assignment Details: All of the 546 patients, 57 (28:XIENCE;29:CYPHER)were excluded from the Per-protocol (PP) population, leaving a baseline population of 489 patients. Whereas because of patient disposition results in a total of 488 patients in the PP population for final analysis.
Period: Overall Study
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Started | 367 | 121
Completed | 360 | 120
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Population: All of the 546 patients, 57 were excluded from the Per-protocol (PP) population, leaving a baseline population of 489 patients and a total of 488 patients (Based on angiographic follow-up) in the PP population for final analysis. In which 367 were randomized to receive XIENCE V EECSS and 121 to CYPHER SELECT Plus SECSS group.
Groups:
- Total: Total of all reporting groups
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS | Total
Number analyzed (Participants) | 367 | 121 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.60 (10.65) | 58.74 (9.12) | 58.64 (10.28)
Age, Customized [Number; unit: participants]
  Age ≥ 65 years | 95 | 33 | 128
  Age < 65 years | 272 | 88 | 360
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 40 | 135
  Male | 272 | 81 | 353
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 367 | 121 | 488
Region of Enrollment [Number; unit: participants]
  China | 367 | 121 | 488

OUTCOME MEASURES:

1. Primary Outcome: In-stent Late Loss (LL)
Description: This is the primary angiographic endpoint.
  In-stent LL: The difference between the minimum lumen diameter (MLD) immediately after stent deployment and the MLD at follow-up (within stent)
Time Frame: >=13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 279 | 98
Number analyzed (Lesions) | 279 | 98
Millimeter | 0.19 (0.28) | 0.21 (0.28)

2. Primary Outcome: Ischemia-driven Target Vessel Failure (ID-TVF)
Description: This is the primary efficacy endpoint. Ischemia-driven target vessel failure is defined as the composite of cardiac death, all myocardial infarction (MI) and ischemia-driven target vessel revascularization (ID-TVR).
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 4.4 [2.51 to 6.98] | 6.6 [2.90 to 12.61]

3. Primary Outcome: Incidence of Composite of ST (Definite and Probable), All Death (Cardiac, Vascular and Non-cardiovascular), and All MI (Including Q-wave and Non-Q-wave)
Description: The primary composite safety endpoint was the incidence of the composite of ST (definite and probable), all death (cardiac, vascular and non-cardiovascular), and all MI (including Q-wave and non-Q-wave).
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.6 [0.60 to 3.52] | 1.7 [0.20 to 5.84]

4. Secondary Outcome: Ischemia-driven Target Vessel Failure (ID-TVF)
Description: Incidence of composite of cardiac death, all MI (including Q-wave and non- Q-wave), and ID target vessel revascularization (ID-TVR) (TLR and non-TLR in the TV [PCI and CABG])
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

5. Secondary Outcome: Ischemia-driven Target Vessel Failure (ID-TVF)
Description: as for outcome 4
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

6. Secondary Outcome: Ischemia-driven Target Vessel Failure (ID-TVF)
Description: as for outcome 4
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.4 | 3.3

7. Secondary Outcome: Ischemia-driven Target Vessel Failure (ID-TVF)
Description: as for outcome 4
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 4.7 | 7.4

8. Secondary Outcome: Incidence of Composite of Stent Thrombosis (ST)(Definite and Probable), All Death (Cardiac, Vascular and Non-cardiovascular), and All MI (Including Q-wave and Non-Q-wave).
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

9. Secondary Outcome: Incidence of Composite of Stent Thrombosis (ST)(Definite and Probable), All Death (Cardiac, Vascular and Non-cardiovascular), and All MI (Including Q-wave and Non-Q-wave).
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

10. Secondary Outcome: Incidence of Composite of Stent Thrombosis (ST)(Definite and Probable), All Death (Cardiac, Vascular and Non-cardiovascular), and All MI (Including Q-wave and Non-Q-wave)
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.4 | 1.7

11. Secondary Outcome: Incidence of Composite of Stent Thrombosis (ST)(Definite and Probable), All Death (Cardiac, Vascular and Non-cardiovascular), and All MI (Including Q-wave and Non-Q-wave)
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 1.9 | 1.7

12. Secondary Outcome: Ischemia-driven Target Lesion Revascularization (ID-TLR) (Percutaneous Coronary Intervention [PCI] and Coronary Artery Bypass Graft [CABG])
Description: The is the major Secondary Efficacy Endpoint.
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.9 [0.77 to 3.89] | 3.3 [0.91 to 8.25]

13. Secondary Outcome: Ischemia-driven Target Lesion Failure (ID-TLF)
Description: Incidence of composite of cardiac death, MI attributed to the TV and ID-TLR
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

14. Secondary Outcome: Ischemia-driven Target Lesion Failure (ID-TLF)
Description: Incidence of composite of cardiac death, MI attributed to the TV and ID-TLR
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

15. Secondary Outcome: Ischemia-driven Target Lesion Failure (ID-TLF)
Description: This is one of the Secondary Composite Endpoints.
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.4 | 2.5

16. Secondary Outcome: Ischemia-driven Target Lesion Failure (ID-TLF)
Description: This is one of the Secondary Composite Endpoints.
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 3.5 | 5.0

17. Secondary Outcome: Ischemia-driven Target Lesion Failure (ID-TLF)
Description: This is one of the Secondary Composite Endpoints.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 3.9 | 5.0

18. Secondary Outcome: Incidence of Composite of Cardiac Death and MI (Including Q-wave and Non-Q-wave) Attributed to the Target Vessel (TV)
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

19. Secondary Outcome: Incidence of Composite of Cardiac Death and MI (Including Q-wave and Non-Q-wave) Attributed to the Target Vessel (TV)
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

20. Secondary Outcome: Incidence of Composite of Cardiac Death and MI (Including Q-wave and Non-Q-wave) Attributed to the Target Vessel (TV)
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.4 | 1.7

21. Secondary Outcome: Incidence of Composite of Cardiac Death and MI (Including Q-wave and Non-Q-wave) Attributed to the Target Vessel (TV)
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.6 | 1.7

22. Secondary Outcome: Incidence of Composite of Cardiac Death and MI (Including Q-wave and Non-Q-wave) Attributed to the Target Vessel (TV)
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 1.7 | 1.7

23. Secondary Outcome: All Death(Cardiac, Vascular and Non-cardiovascular), All MI, All Revascularization (TLR, TVR, and Non-TVR) (PCI and CABG)
Description: This is one of the Secondary Composite Endpoint. All death(cardiac, vascular and non-cardiovascular), all MI, all revascularization [(target lesion revascularization (TLR), target vessel revascularization (TVR), and non-target lesion revascularization(TVR) [Percutaneous coronary intervention (PCI) and Coronary artery bypass graft(CABG)].
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 1.7

24. Secondary Outcome: All Death(Cardiac, Vascular and Non-cardiovascular), All MI, All Revascularization (TLR, TVR, and Non-TVR) (PCI and CABG)
Description: as for outcome 23
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.6 | 2.5

25. Secondary Outcome: All Death(Cardiac, Vascular and Non-cardiovascular), All MI, All Revascularization (TLR, TVR, and Non-TVR) (PCI and CABG)
Description: as for outcome 23
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 2.2 | 5.0

26. Secondary Outcome: All Death(Cardiac, Vascular and Non-cardiovascular), All MI, All Revascularization (TLR, TVR, and Non-TVR) (PCI and CABG)
Description: as for outcome 23
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 6.3 | 10.7

27. Secondary Outcome: All Death(Cardiac, Vascular and Non-cardiovascular), All MI, All Revascularization (TLR, TVR, and Non-TVR) (PCI and CABG)
Description: as for outcome 23
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 8.5 | 11.6

28. Secondary Outcome: Incidence of Composite of All Death (Cardiac, Vascular and Non-cardiovascular) and All MI
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

29. Secondary Outcome: Incidence of Composite of All Death (Cardiac, Vascular and Non-cardiovascular) and All MI
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

30. Secondary Outcome: Incidence of Composite of All Death (Cardiac, Vascular and Non-cardiovascular) and All MI
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.4 | 1.7

31. Secondary Outcome: Incidence of Composite of All Death (Cardiac, Vascular and Non-cardiovascular) and All MI
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.6 | 1.7

32. Secondary Outcome: Incidence of Composite of All Death (Cardiac, Vascular and Non-cardiovascular) and All MI
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 1.9 | 1.7

33. Secondary Outcome: Major Adverse Cardiac Event (Cardiac Death, All MI and TLR)
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

34. Secondary Outcome: Major Adverse Cardiac Event (Cardiac Death, All MI and TLR)
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

35. Secondary Outcome: Major Adverse Cardiac Event (Cardiac Death, All MI and TLR)
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.4 | 2.5

36. Secondary Outcome: Major Adverse Cardiac Event (Cardiac Death, All MI and TLR)
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 3.5 | 5.0

37. Secondary Outcome: Major Adverse Cardiac Event (Cardiac Death, All MI and TLR)
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 3.9 | 5.0

38. Secondary Outcome: All Revascularization (TLR, TVR, and Non-TVR)
Time Frame: 30 Days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.3 | 0.8

39. Secondary Outcome: All Revascularization (TLR, TVR, and Non-TVR)
Time Frame: 6 Months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.5 | 1.7

40. Secondary Outcome: All Revascularization (TLR, TVR, and Non-TVR)
Time Frame: 9 Months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 3.3

41. Secondary Outcome: All Revascularization (TLR, TVR, and Non-TVR)
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 4.6 | 9.1

42. Secondary Outcome: All Revascularization (TLR, TVR, and Non-TVR)
Description: One of the Secondary Safety Endpoint was all revascularization rates (target lesion, target vessel, non-target lesion, and non-target vessel) (PCI and CABG).
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 6.6 | 9.9

43. Secondary Outcome: All Death
Description: This is one of the secondary safety endpoint. All Death includes cardiac, vascular, non-cardiovascular.
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.0 | 0.0

44. Secondary Outcome: All Death
Description: This is one of the secondary safety endpoint. All Death includes cardiac, vascular, non-cardiovascular.
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.3 | 0.0

45. Secondary Outcome: All Death
Description: This is one of the secondary safety endpoint. All Death includes cardiac, vascular, non-cardiovascular.
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.5 | 0.8

46. Secondary Outcome: All Death
Description: This is one of the secondary safety endpoint. All Death includes cardiac, vascular, non-cardiovascular.
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.5 | 0.8

47. Secondary Outcome: All Death
Description: This is one of the secondary safety endpoint. All Death includes cardiac, vascular, non-cardiovascular.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 0.8 | 0.8

48. Secondary Outcome: All Protocol MI (Including Q-wave or Non-Q-wave)
Description: This is one of the secondary safety endpoint.
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

49. Secondary Outcome: All Protocol MI (Including Q-wave or Non-Q-wave)
Description: This is one of the secondary safety endpoint.
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

50. Secondary Outcome: All Protocol MI (Including Q-wave or Non-Q-wave)
Description: This is one of the secondary safety endpoint.
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

51. Secondary Outcome: All Protocol MI (Including Q-wave or Non-Q-wave)
Description: This is one of the secondary safety endpoint.
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

52. Secondary Outcome: All Protocol MI (Including Q-wave or Non-Q-wave)
Description: This is one of the secondary safety endpoint.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 1.1 | 0.8

53. Secondary Outcome: Target Vessel Protocol MI (TV-MI)
Description: This is one of the secondary safety endpoint.
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

54. Secondary Outcome: Target Vessel Protocol MI (TV-MI)
Description: This is one of the secondary safety endpoint.
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

55. Secondary Outcome: Target Vessel Protocol MI (TV-MI)
Description: This is one of the secondary safety endpoint.
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.8 | 0.8

56. Secondary Outcome: Target Vessel Protocol MI (TV-MI)
Description: This is one of the secondary safety endpoint.
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 1.1 | 0.8

57. Secondary Outcome: Target Vessel Protocol MI (TV-MI)
Description: This is one of the secondary safety endpoint.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 363 | 121
percentage of participants | 1.1 | 0.8

58. Secondary Outcome: Major Bleeding Complications
Description: Secondary safety endpoint.
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.0 | 0.0

59. Secondary Outcome: Major Bleeding Complications
Description: Secondary safety endpoint.
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.0 | 0.0

60. Secondary Outcome: Major Bleeding Complications
Description: Secondary safety endpoint.
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 366 | 121
percentage of participants | 0.0 | 0.0

61. Secondary Outcome: Major Bleeding Complications
Description: Secondary safety endpoint.
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 365 | 121
percentage of participants | 0.5 | 0.0

62. Secondary Outcome: Major Bleeding Complications
Description: Secondary safety endpoint.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 360 | 120
percentage of participants | 0.8 | 0.0

63. Secondary Outcome: Definite / Probable Stent Thrombosis
Description: Stent Thrombosis was adjudicated using Academic Research Consortium (ARC) criteria. Definite Stent Thrombosis defined as angiographic confirmation with at least one of the following: acute onset of ischemic symptoms at rest, new ischemic changes suggestive of acute ischemia, typical rise and fall of cardiac biomarkers; pathological confirmation of ST through either autopsy or tissue examination following thrombectomy. Probable Stent Thrombosis defined as any unexplained death within the first 30 days or, irrespective of the time after the index procedure, any MI related to documented acute ischemia in the territory of the stent without angiographic confirmation.
Time Frame: Acute (<1 day)
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.27 | 0.00

64. Secondary Outcome: Definite / Probable Stent Thrombosis
Description: as for outcome 63
Time Frame: Subacute (1 - 30 days)
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.27 | 0.00

65. Secondary Outcome: Definite / Probable Stent Thrombosis
Description: as for outcome 63
Time Frame: Early (0 - 30 days)
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.54 | 0.00

66. Secondary Outcome: Definite / Probable Stent Thrombosis
Description: as for outcome 63
Time Frame: Late (31 - 365 days)
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.00 | 0.00

67. Secondary Outcome: Definite / Probable Stent Thrombosis
Description: as for outcome 63
Time Frame: Very late (366 - 772 days)
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.00 | 0.00

68. Secondary Outcome: Definite / Probable Stent Thrombosis
Description: as for outcome 63
Time Frame: Overall (0 - 772 days)
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 0.54 | 0.00

69. Secondary Outcome: Patient Compliance With Dual Antiplatelet Therapy (DAPT)
Time Frame: 30 days
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 362 | 121
percentage of participants | 99.2 | 99.2

70. Secondary Outcome: Patient Compliance With Dual Antiplatelet Therapy (DAPT)
Time Frame: 6 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 362 | 121
percentage of participants | 99.2 | 97.5

71. Secondary Outcome: Patient Compliance With Dual Antiplatelet Therapy (DAPT)
Time Frame: 9 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 362 | 121
percentage of participants | 98.1 | 95.9

72. Secondary Outcome: Patient Compliance With Dual Antiplatelet Therapy (DAPT)
Time Frame: 12 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 362 | 121
percentage of participants | 94.5 | 93.4

73. Secondary Outcome: Patient Compliance With Dual Antiplatelet Therapy (DAPT)
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 362 | 121
percentage of participants | 58.0 | 55.4

74. Secondary Outcome: Acute Device Success
Description: Per-protocol device success is defined as the achievement of a final in-stent residual diameter stenosis (DS) of < 50% by Quantitative Coronary Angiography (QCA), using only the assigned device, and occurring without a device malfunction.
Time Frame: < or = 1 day
Measure: Number; unit: percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Number analyzed (Target lesions) | 399 | 129
percentage of participants | 97.2 | 98.4

75. Secondary Outcome: Acute Procedure Success
Description: Per-protocol procedure success is defined as the achievement of a final in-stent DS of < 50% (by online QCA or visual estimation), using the assigned device and with any adjunctive devices, and occurring without cardiac death, MI (including Q-wave or non-Q-wave), or repeat revascularization of the target lesion during the hospital stay.
Time Frame: < or = 1 day
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
percentage of participants | 98.1 | 99.2

76. Secondary Outcome: Procedure Time
Description: This is the procedure related endpoint. Procedure time is defined as time between insertion of the first guiding catheter until removal of the last guiding catheter.
Time Frame: On day 0, during the procedure.
Measure: Median (Standard Deviation); unit: Minutes
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Minutes | 29.6 (19.3) | 28.6 (15.8)

77. Secondary Outcome: Amount of Contrast Used
Description: Defined as total amount used from insertion of the first guiding catheter until removal of the last guiding catheter.
Time Frame: On day 0, during the procedure.
Measure: Median (Standard Deviation); unit: Milliliter
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Milliliter | 132.1 (53.2) | 145.4 (59.2)

78. Secondary Outcome: Fluoroscopy Time
Description: This is the procedure related endpoint.
Time Frame: On day 0, during the procedure.
Measure: Median (Standard Deviation); unit: Minutes
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Minutes | 7.0 (4.7) | 7.4 (4.7)

79. Secondary Outcome: XIENCE V EECSS Excellent Overall Performance and Deliverability Using the XIENCE V EECSS Performance Evaluation Questionnaire
Description: A related secondary performance goal for XIENCE V EECSS is the physician-determined evaluation of acute performance, deliverability, and resource utilization. XIENCE V EECSS acute performance and deliverability were determined using the XIENCE V EECSS Performance Evaluation Questionnaire. Possible responses included strongly agree,moderately agree, agree, moderately disagree, and strongly disagree. Study physicians who enrolled patients into the study were reported for this outcome measure.
Time Frame: During the procedure
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS
Number analyzed (Participants) | 367
percentage of participants | 93.2

80. Secondary Outcome: Follow-up Late Loss
Description: This is one of the Secondary Angiographic Endpoint.
Time Frame: ≥13 months.
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 279 | 98
Number analyzed (Target lesions) | 279 | 98
Millimeter
  In-Segment | 0.15 (0.35) | 0.27 (0.35)
  Proximal | 0.20 (0.34) | 0.33 (0.39)
  Distal | 0.11 (0.32) | 0.20 (0.33)

81. Secondary Outcome: Follow-up In-stent Minimum Lumen Diameter (MLD)
Time Frame: ≥13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 280 | 98
Number analyzed (Target lesions) | 280 | 98
Millimeter | 2.62 (0.50) | 2.63 (0.48)

82. Secondary Outcome: Follow-up In-stent Percent Diameter Stenosis (DS)
Time Frame: ≥13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 280 | 98
Number analyzed (Target lesions) | 280 | 98
percent Diameter stenosis | 10.56 (10.18) | 11.82 (10.30)

83. Secondary Outcome: Follow-up In-stent Angiographic Binary Restenosis (ABR)
Time Frame: ≥13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 280 | 98
Number analyzed (Target lesions) | 280 | 98
percentage of participants | 1.1 | 1.0

84. Secondary Outcome: Follow-up In-segment Minimum Lumen Diameter (MLD)
Time Frame: ≥13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 280 | 98
Number analyzed (Target lesions) | 280 | 98
Millimeter | 2.34 (0.52) | 2.33 (0.50)

85. Secondary Outcome: Follow-up In-segment Percent Diameter Stenosis (DS)
Time Frame: ≥13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 280 | 98
Number analyzed (Target lesions) | 280 | 98
percent Diameter stenosis | 16.79 (12.36) | 18.79 (12.42)

86. Secondary Outcome: Follow-up In-segment Angiographic Binary Restenosis (ABR)
Time Frame: ≥13 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 280 | 98
Number analyzed (Target lesions) | 280 | 98
percentage of participants | 2.1 | 3.1

87. Secondary Outcome: Percent Diameter Stenosis
Time Frame: pre procedure
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Number analyzed (Target lesions) | 398 | 129
percent Diameter stenosis | 64.97 (11.90) | 64.95 (12.01)

88. Secondary Outcome: Percent Diameter Stenosis (%DS)
Time Frame: post procedure on 0 day
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Number analyzed (Target lesions) | 398 | 129
Percent Diameter stenosis
  in-stent %DS | 8.09 (6.31) | 8.56 (5.78)
  in-segment %DS | 14.40 (8.09) | 12.46 (7.41)

89. Secondary Outcome: Acute Gain
Time Frame: post procedure on 0 day
Population: The number of participants with angiographic follow up available was analysed.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Target lesions
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 367 | 121
Number analyzed (Target lesions) | 398 | 129
Millimeter
  In-Stent | 1.79 (0.44) | 1.77 (0.43)
  In-Segment | 1.48 (0.49) | 1.52 (0.44)
  Proximal | 2.03 (0.53) | 2.06 (0.49)
  Distal | 1.54 (0.54) | 1.60 (0.51)

90. Other Pre Specified Outcome: ID-TVF Rate in Patients With Diabetic Disease
Description: ID-TVF rate in All Diabetes patients.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 87 | 29
percentage of participants | 5.7 | 13.8

91. Other Pre Specified Outcome: ID-TVF Rate in Patients Without Diabetic Disease
Description: ID-TVF rate in Non Diabetes
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 272 | 91
percentage of participants | 4.4 | 5.5

92. Other Pre Specified Outcome: ID-TVF Rate in Single Lesion Treated Subgroup
Description: ID-TVF rate in Patients with single lesion treated during the index procedure
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 332 | 113
percentage of participants | 4.8 | 7.1

93. Other Pre Specified Outcome: ID-TVF Rate in Dual Lesion Treated Subgroup
Description: ID-TVF rate in Patients with dual lesion treated during the index procedure
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 30 | 8
percentage of participants | 3.3 | 12.5

94. Other Pre Specified Outcome: ID-TVF Rate in Single Vessel Treated Subgroup
Description: ID-TVF rate in Patients with single vessels treated during the index procedure.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 339 | 114
percentage of participants | 4.7 | 7.0

95. Other Pre Specified Outcome: ID-TVF Rate in Dual Vessel Treated Subgroup
Description: ID-TVF rate in Patients with dual vessel treated during the index procedure.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 24 | 7
percentage of participants | 4.2 | 14.3

96. Other Pre Specified Outcome: The Composite of ST, All Death, and All MI Rate in Patients With Diabetic Disease.
Description: The composite of ST, all death, and all MI rate in All Diabetes patients.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 87 | 29
percentage of participants | 1.1 | 3.4

97. Other Pre Specified Outcome: The Composite of ST, All Death, and All MI Rate in Patients Without Diabetic Disease
Description: The composite of ST, all death, and all MI rate in Non Diabetes
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 272 | 91
percentage of participants | 2.2 | 1.1

98. Other Pre Specified Outcome: The Composite of ST, All Death, and All MI Rate in Single Lesion Treated Subgroup
Description: The composite of ST, all death, and all MI rate in Patients with single lesion treated during the index procedure
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 332 | 113
percentage of participants | 1.8 | 1.8

99. Other Pre Specified Outcome: The Composite of ST, All Death, and All MI Rate in Dual Lesion Treated Subgroup
Description: The composite of ST, all death, and all MI rate in Patients with dual lesion treated during the index procedure
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 30 | 8
percentage of participants | 3.3 | 0.0

100. Other Pre Specified Outcome: The Composite of ST, All Death, and All MI Rate in Single Vessel Treated Subgroup
Description: The composite of ST, all death, and all MI rate in Patients with single vessels treated during the index procedure.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 339 | 114
percentage of participants | 1.8 | 1.8

101. Other Pre Specified Outcome: The Composite of ST, All Death, and All MI Rate in Dual Vessel Treated Subgroup
Description: The composite of ST, all death, and all MI rate in Patients with dual vessel treated during the index procedure.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 24 | 7
percentage of participants | 4.2 | 0.0

102. Other Pre Specified Outcome: ID-TLR Rate in Patients With Diabetic Disease.
Description: Ischemia-driven target lesion revascularization rate in All Diabetes patients.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 87 | 29
percentage of participants | 3.4 | 3.4

103. Other Pre Specified Outcome: ID-TLR Rate in Patients Without Diabetic Disease
Description: Ischemia-driven target lesion revascularization rate in Non Diabetes
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 272 | 91
percentage of participants | 1.8 | 3.3

104. Other Pre Specified Outcome: ID-TLR Rate in Single Lesion Treated Subgroup
Description: Ischemia-driven target lesion revascularization rate in Patients with single lesion treated during the index procedure
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 332 | 113
percentage of participants | 2.4 | 2.7

105. Other Pre Specified Outcome: ID-TLR Rate in Dual Lesion Treated Subgroup
Description: Ischemia-driven target lesion revascularization rate in Patients with dual lesion treated during the index procedure
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 30 | 8
percentage of participants | 0.00 | 12.5

106. Other Pre Specified Outcome: ID-TLR Rate in Single Vessel Treated Subgroup
Description: Ischemia-driven target lesion revascularization rate in Patients with single vessels treated during the index procedure.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 339 | 114
percentage of participants | 2.4 | 2.6

107. Other Pre Specified Outcome: ID-TLR Rate in Dual Vessel Treated Subgroup
Description: Ischemia-driven target lesion revascularization rate in Patients with dual vessel treated during the index procedure.
Time Frame: 24 months
Population: The number of participants with angiographic follow up available was analysed.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Number analyzed (Participants) | 24 | 7
percentage of participants | 0.0 | 14.3

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | XIENCE V EECSS | CYPHER SELECT PLUS SECSS
Serious Adverse Events (participants affected / at risk) | 53/360 | 24/120
Other Adverse Events (participants affected / at risk) | 32/360 | 14/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE V EECSS (N=360) | CYPHER SELECT PLUS SECSS (N=120)
Angina (Cardiac disorders) | 7 (8) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block (AVB) (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 3 (3) | 1 (1)
Creatine kinase MB (CK-MB) increased (Investigations) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Dissection (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Heart Disease (Cardiac disorders) | 1 (1) | 1 (1)
Death (General disorders) | 3 (3) | 0 (0)
Fibrillation Atrial (Cardiac disorders) | 2 (2) | 0 (0)
Gastric Ulcer With Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hear Failure (Cardiac disorders) | 1 (1) | 2 (3)
Melena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Non-Targeted Vessel Revascularization (Surgical and medical procedures) | 1 (1) | 0 (0)
Restenosis (Surgical and medical procedures) | 3 (3) | 3 (4)
Revascularization (Surgical and medical procedures) | 9 (9) | 0 (0)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Target Lesion Revascularization (Surgical and medical procedures) | 2 (2) | 1 (1)
Non-Target Vascular Stenosis (Surgical and medical procedures) | 2 (2) | 0 (0)
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Respiratory Fail, Chronic Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Unstable Angina (Cardiac disorders) | 4 (5) | 3 (3)
Upper Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vascular Stenosis (Vascular disorders) | 1 (1) | 1 (1)
Extrasystole; Fibrillation Atrial (Cardiac disorders) | 0 (0) | 1 (2)
Coronary heart disease (CHD), Coronary Revascularization (Cardiac disorders) | 0 (0) | 1 (1)
Liver Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (3)
Target Vessel Revasculization (Surgical and medical procedures) | 0 (0) | 1 (1)
Non-Target Vessel Restenosis (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XIENCE V EECSS (N=360) | CYPHER SELECT PLUS SECSS (N=120)
Angina (Cardiac disorders) | 1 (1) | 1 (1)
Chest Distress Because Of Air Pollution (General disorders) | 1 (1) | 0 (0)
Chest Distress Occasionally (General disorders) | 1 (1) | 1 (1)
Chest Pain Happens More Frequently (General disorders) | 1 (1) | 0 (0)
Chest Tightness (General disorders) | 1 (1) | 1 (1)
Creatine kinase-MB (CK-MB0 Increase (Investigations) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac troponin T increased (cTnI) (Investigations) | 6 (6) | 2 (2)
Cardiac troponin T of Post-Procedure Increased (Investigations) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (MI) (Cardiac disorders) | 1 (1) | 0 (0)
Peri-procedural PCI and MI (Surgical and medical procedures) | 2 (2) | 0 (0) — Peri-procedural percutaneous coronary intervention (PCI) and peri-procedural myocardial infarction
Premature Beat (General disorders) | 1 (1) | 0 (0)
The Cardiac Enzyme Is Higher (Investigations) | 1 (1) | 0 (0)
Abnormal troponin I (TnI) (Investigations) | 1 (1) | 0 (0)
Troponin I (TnI) Increase (Investigations) | 5 (5) | 2 (2)
Troponin I (TnI) Increase Significantly (Investigations) | 2 (2) | 1 (1)
Troponin I (TnI) Of Post Procedure Increased (Investigations) | 2 (2) | 2 (2)
Troponin T (TnT) of Post Procedure Increased (Investigations) | 1 (1) | 0 (0)
Vessel Interlayer (Surgical and medical procedures) | 1 (1) | 0 (0)
Breathing Difficulty (General disorders) | 0 (0) | 1 (1)
Complication of percutaneous coronary intervention (PCI) Procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrorrhagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasal Bleeding (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No